CLINICAL TRIAL: NCT00108147
Title: Functional Circuit Training in Older Adults With Congestive Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Alexander, Neil - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: AGCG-002-03S
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Heart Failure, Congestive
Keywords: Aged; Congestive Heart Failure; Exercise
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Circuit-Based Exercise; Cardiac Rehabilitation; Pliability

ARMS (3):
- 1 (Experimental): Circuit Training
  Interventions: Procedure: Circuit Training
- 2 (Active Comparator): Cardiac Rehabilitation
  Interventions: Procedure: Cardiac Rehabilitation
- 3 (Active Comparator): Flexibility and toning
  Interventions: Procedure: Flexibility and toning

INTERVENTIONS:
Procedure: Circuit Training
  Arms: 1
Procedure: Cardiac Rehabilitation
  Arms: 2
Procedure: Flexibility and toning
  Arms: 3

SUMMARY:
The goal of this study is to determine the effect of a functional circuit training program as compared to standard cardiac rehabilitation or control exercise in improving physical function and activity.

DETAILED DESCRIPTION:
In older (65 years of age or older) patients with congestive heart failure, we propose to:

1. Assess: a) Peak aerobic capacity (peak VO2) during a monitored, standardized treadmill test; b) Oxygen uptake kinetics and heart rate during a standardized submaximal treadmill test; c) Performance on a set of functional mobility tasks; d) Self-report of physical disability and difficulty in performing daily tasks, and physical activity.
2. Conduct a 12-week randomized controlled trial, comparing changes in these assessed measures in patients randomized to three different groups: 1) standard cardiac rehabilitation using bicycle exercise; 2) group functional circuit training focusing on exercises that involve functional mobility tasks and a home-activities exercise component; 3) a chair-based, flexibility and "toning " (low level resistance) group control exercise.
3. Reassess all groups after an additional 12 weeks in the measures identified above to identify how well the three groups maintain their function.
4. Examine the mechanisms underlying change in functional mobility performance and self-reported function as a result of the interventions

Primary hypothesis 1: Compared to chair-based exercise controls at the end of week 12, both the cardiac rehabilitation and functional circuit training groups will show improvements in measures of peak aerobic capacity, submaximal oxygen uptake kinetics, functional mobility performance, and self-reported function.

Primary hypothesis 2: Compared to the other two groups that are given exercise instructions only, the functional circuit training group, who continue their home activities exercise program, show less decline by week 24 in measures of peak aerobic capacity, submaximal oxygen uptake kinetics, functional mobility performance, and self-reported function.

Secondary hypothesis: Measures of submaximal oxygen uptake kinetics are better predictors of changes in functional mobility performance and self-reported function than peak aerobic capacity, muscle strength, joint range of motion, balance, and behavioral factors (such as depression).

ELIGIBILITY:
Inclusion Criteria:

* Congestive Heart Failure

Exclusion Criteria:

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10

CONTACTS AND LOCATIONS:
Overall Officials: Neil Alexander, MD, Principal Investigator — VA Ann Arbor Healthcare System
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States